CLINICAL TRIAL: NCT00254761
Title: A Double Blind, Active Placebo Controlled Crossover Trial of the Antinociceptive Effect of Smoked Marijuana on Subjects With Neuropathic Pain; Correlation With Changes in Mood, Cognition, and Psychomotor Performance
Brief Title: Effects of Smoked Marijuana on Neuropathic Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Center for Medicinal Cannabis Research (Other)
Responsible Party: Barth Wilsey, M.D., University of California, Davis
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C02-DA-114
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Neuropathic Pain
Keywords: cannabis; marijuana; neuropathy; antinociception; mood; cognition
MeSH Terms: conditions — Neuralgia; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): High dose cannabis (7.5% THC by weight)
  Interventions: Drug: Cannabis
- 2 (Experimental): Low dose cannabis (3.5% THC by weight)
  Interventions: Drug: Cannabis
- 3 (Placebo Comparator): Placebo cannabis
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis

SUMMARY:
To determine if smoking marijuana will reduce neuropathic pain without causing too much drowsiness or feeling "too dopey".

DETAILED DESCRIPTION:
The case for marijuana's medical use for pain is primarily from experimental studies with normal subjects, which have yielded conflicting results. Experimental subjects have been shown to have significant dose-dependant antinociception effect that is not reversed by opioid antagonism. In contrast to this positive antinociceptive effect, other experiments demonstrated hyperalgesic activity and probably enhancement of the perception of pain upon acute exposure in chronic users of marijuana.

In addition to studying spontaneous pain antinociception, it would be useful to evaluate the response to marijuana following evoked pain. Such evoked pain is produced by stimulation of the skin that is normally not noxious.

Because of the potential side effects of marijuana administration, one of the aims of the present study is to analyze inter-individual variability and the occurrence of dose-dependant analgesia of marijuana with an eye on defining tolerable dosing in clinical neuropathic pain syndromes.

Comparisons: Neuropathic and experimentally induced pain scores will be compared after the administration of escalating doses of low, high, and placebo marijuana cigarettes as provided by the National Institutes on Drug Abuse (NIDA).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand English
* Age greater than 18 and less than 70
* VAS greater than 3/10
* History of previous marijuana use (i.e., avoidance of marijuana naive subjects)
* Negative urine drug screening test
* Nerve Injury a.k.a. Complex Regional Pain Syndrome Type II OR
* Complex Regional Pain Syndrome Type I OR
* Neuropathic pain due to confirmed bilateral distal peripheral neuropathy associated with Diabetes I or II, focal nerve injury, postherpetic neuralgia, spinal cord injury with incomplete myelopathy, central pain following a stroke or focal brain lesion, or clinical definite multiple sclerosis of at least 3 months duration.

Exclusion Criteria:

* Presence of another painful condition of greater severity than the neuropathic pain condition which is being studied
* Unstable Type 1 or 2 diabetes defined as blood glucose more than 156 mg/dl
* For diabetic subjects maintained on insulin with a stable blood glucose more than 156 mg/dl, a hemoglobin A1C level of more than 0.11 (normal range, 0.048-0.067)
* History of traumatic brain injury
* History of schizophrenia or a past or current history of a serious psychiatric disorder that is currently not well controlled with medications
* Uncontrolled medical condition - coronary artery disease, hypertension, cerebrovascular disease, asthma, TB, COPD, opportunistic infection, malignancy requiring active treatment
* Active substance abuse (alcohol or injection drugs)
* Current use of marijuana (within 30 days of randomization) as determined by urine screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Score on a series of pain scales (heat pain threshold, VAS intensity, VAS unpleasantness, pain relief, neuropathic pain scale).

SECONDARY OUTCOMES:
Number of subjects who are unable to tolerate the high dose without significant side effects.
Changes in mood, cognitive impairment, and psychomotor performance (mood - VAS happiness, cognition - Digit Symbol Modalities Test, psychomotor performance - Grooved Pegboard Test).

CONTACTS AND LOCATIONS:
Overall Officials: Barth L Wilsey, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- See also: Center For Medicinal Cannabis Research — http://cmcr.ucsd.edu